CLINICAL TRIAL: NCT00381979
Title: Supportive Expressive Therapy for Depressed and Anxious Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Pamela Wilansky-Traynor, psychologist, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 169/2003
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-09

CONDITIONS: Depression; Anxiety
Keywords: Depression; Anxiety; Adolescents; Treatment; Supportive Expressive Therapy
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): set
  Interventions: Other: Supportive Expressive Therapy

INTERVENTIONS:
Other: Supportive Expressive Therapy
  Other Names: therapy

SUMMARY:
The purpose of the study is to investigate the effectiveness of providing Supportive Expressive Therapy to adolescents who are depressed and/or anxious.

DETAILED DESCRIPTION:
Supportive Expressive Therapy (SET; a 16 session manualized form of psychodynamic therapy) has been well utilized with adult clients. To date, there is no known systematic study into the benefit of this method of therapy with adolescents who are depressed and/or anxious. It is thought that SET would be useful for this population as it is similar in principle to Interpersonal Relationship Therapy (IPT), which has been shown to be effective for use with depressed adults and youth. Both IPT and SET help clients explore the role they play within challenging relationships in their lives. SET, however, allows for the exploration of more relationships within the adolescents' circle. Moreover, SET explores the adolescents' perceptions of themselves, others, and their wish in relationships. Further, the SET method is more easily individualized in that it affords greater flexibility in design and possibility for change over time. Accordingly, the purpose of this study is to explore the feasibility of utilizing this method of therapy with adolescents who are depressed and anxious. We will be exploring the effectiveness of SET through the resolution of depressed and/or anxious adolescents' conflictual relationships thereby reducing their symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* 15-24 year old, male & female adolescents, primary diagnosis of depression or anxiety disorder.
* Clients with co-morbid diagnoses, suicidal ideation or taking medication would not necessarily be excluded if deemed able to partake in the proposed therapy.
* Medication dose needs to be stable for 4-6 weeks prior to starting therapy.

Exclusion Criteria:

* Clients who are actively psychotic, developmentally delayed, or have a diagnosis of bipolar disorder.
* Clients who are not fluent in English.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2004-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
BDI | pre and post
MASC | pre and post
Measures collected at pre, post, and follow-up | pre and post

SECONDARY OUTCOMES:
YSR | pre and post
CBCL | pre and post
FAM | pre and post
CRI | pre and post
SSRS | pre and post
Measures collected at pre, post, and follow-up | pre and post

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada